CLINICAL TRIAL: NCT05881785
Title: A Randomized, Double-blind, Placebo-controlled, Phase III Study of Efficacy and Safety of GR1501 in Patients with Radiographic Axial Spondyloarthritis
Brief Title: Study of Efficacy and Safety of GR1501 in Patients with Radiographic Axial Spondyloarthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genrix (Shanghai) Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GR1501-007
Record Dates: First submitted 2023-05-21; First posted 2023-05-31 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Axial Spondyloarthritis
Keywords: IL-17A; Autoimmune disease
MeSH Terms: conditions — Axial Spondyloarthritis; Autoimmune Diseases

STUDY DESIGN:
Intervention Model Description: A total of 465 patients were randomly assigned to 100mg GR1501 injection, 200mg GR1501 injection, and placebo group at 1:1:1. Randomized stratification factors included history of biologic therapy and weight. After the completion of 16-week ,subjects in the GR1501 injection group continued to be administered GR1501 injection, and those in the placebo group were randomly assigned 1:1 to the 100mg GR1501 injection and 200mg GR1501 injection.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Treatment group 1 (Experimental): GR1501 low dose
  Interventions: Biological: GR1501 low dose
- Treatment group 2 (Experimental): GR1501 high dose
  Interventions: Biological: GR1501 high dose
- treatment group 3 (Placebo Comparator): placebo
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: GR1501 low dose — 3×low dose GR1501 every 2 weeks,then low dose GR1501 monthly
  Arms: Treatment group 1
Biological: GR1501 high dose — 3×high dose GR1501 every 2 weeks,then high dose GR1501 monthly
  Arms: Treatment group 2
Biological: placebo — * Core treatment period:placebo
  * Maintenance treatment period: GR1501 injection
  Arms: treatment group 3

SUMMARY:
The purpose of this trial is to demonstrate the clinical efficacy of GR1501 at week 16; and to demonstrate safety and tolerability of GR1501 compared to placebo in patients with Radiographic Axial Spondyloarthritis at week 16 and long term safety up to Week 48。 The main question it aims to answer is whether GR1501 injection was superior to placebo in the proportion of subjects with ASAS20 response at week 16 in patients with Radiographic Axial Spondyloarthritis.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, multicenter clinical study to evaluate the efficacy and safety of GR1501 injection in Radiographic Axial Spondyloarthritis, as well as a confirmatory clinical trial of immunogenicity.

This clinical trial was divided into four stages, namely screening period (W-4~W0), core treatment period (W0~W16), maintenance treatment period (W16~W32), and follow-up period (W32~W48).

target population： radiographic axial spondyloarthritis who had a inadequate response to NSAIDs or have a history of intolerance to NSAIDs.

primary outcome measure:percentage of participants achieving an ASAS20 response in week 16.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of radiographic axial spondyloarthritis (r-xSpA) with sacroiliitis defined radiographically according to the modified New York criteria.
* inadequate response, contraindications or intolerance to NSAIDs

Exclusion Criteria:

* Total ankylosis of the spine
* Ongoing or serious infection
* Either a current diagnosis or a recent history of malignant disease
* Are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 465 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2024-05-21 (Actual)

PRIMARY OUTCOMES:
The Proportion of Participants Who Achieve an ASAS 20 Response | week 16
  ASAS20 response is defined as an improvement of ≥20% and ≥1 units in at least three of the four ASAS main domains

SECONDARY OUTCOMES:
The Proportion of Participants Who Achieve an ASAS 20 Response | week 2 to 48
  ASAS20 response is defined as an improvement of ≥20% and ≥1 units in at least three of the four ASAS main domains
The Proportion of Participants Who Achieve an ASAS 40 Response | week 2 to 48
  ASAS40 response is defined as an improvement of ≥40% and ≥2 units in at least three of the four ASAS main domains
The Proportion of Participants Who Achieve an ASAS 5/6 Response | week 16，32，48
  The ASAS 5/6 improvement criteria is an improvement of ≥20% in at least five of all six domains
Change From Baseline in Mobility on the BASMI | week 16，32，48
  5 clinical measurements Bath Ankylosing Spondylitis Metrology Index
Change From Baseline in BASDAI Response | week 16，32，48
  6 questions that relate to 5 major symptoms relevant to radiographic axial spondyloarthritis
Change From Baseline in Bath Ankylosing Spondylitis Functional Index (BASFI) | week 16，32，48
  10 questions to assess the disease severity, including the first 8 questions regarding to functional anatomy related activities and the remaining 2 questions related to daily activities
Change From Baseline in Maastricht Ankylosing Spondylitis Enthesitis Score (MASES) | week 16，32，48
  The MASES assesses 13 sites for enthesitis using a score of "0" for no activity or "1" for activity
Change From Baseline in Ankylosing Spondylitis Disease Activity Score (ASDAS) | week 16，32，48
  ASDAS is a composite index to assess disease activity in AS

CONTACTS AND LOCATIONS:
Overall Officials: xiaofeng zeng, PHD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking union Medical Hosipital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang S, Xu D, Liu S, Li S, Wang X, Yuan F, Gou W, Xu B, Sun L, Gu J, Zhou D, Li X, Kong N, Zhao Y, Hao J, Li T, Fan X, Shu Q, Wei H, Jiang T, Yang J, Qian L, Sun H, Cai X, Jiang Z, Yuan G, Qin L, Yang M, Xu J, Fan W, Sun L, Zhang H, Zhang C, Zhang N, Da Z, Hu J, Jin J, Liu J, Dai L, Dong L, Wang W, Zeng X. Xeligekimab, an Interleukin-17A Antagonist for Active Radiographic Axial Spondyloarthritis in Chinese Patients: 16- and 48-Week Results from a Phase III, Randomized, Double-Blind, Placebo-Controlled Study. BioDrugs. 2026 Jan;40(1):151-162. doi: 10.1007/s40259-025-00750-0. Epub 2025 Nov 17. PMID 41247398